CLINICAL TRIAL: NCT03597958
Title: Genetic Causes of Hypercholesterolaemia in the Emirati Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London Diabetes Centre (Other)
Responsible Party: Sponsor
Other Study IDs: IREC027
Record Dates: First submitted 2018-06-27; First posted 2018-07-24 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-02

CONDITIONS: Familial Hypercholesterolemia
Keywords: Familial Hypercholesterolemia; Hypercholesterolemia; Cascade Screening; Novel FH Genes; Novel FH Mutations; Next generation sequencing
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA will be extracted from collected blood samples for genetic analysis

GROUPS / COHORTS (1):
- Hypercholesterolaemia: Individuals attending Imperial College London Diabetes Centre (ICLDC) and with LDL-C ≥5.0 mmol/L, for children <18 years LDL-C>95th centile by age and gender for country, and possible evidence of known premature CHD.
  Individuals with a high probability of disease according to the Dutch Lipid Network Criteria, score of ≥6 points, will be identified as possible probands (individual serving as our starting point for the genetic study of the family) and will be selected for further screening.
  Patients will be tested for known and/or suspected FH genes, using next generation sequencing (NGS) panel, whole exome and/or whole genome sequencing (WES/WGS) in cases where FH is highly suspected despite negative results from panel testing, and transcriptomic analysis of RNA blood samples.
  Interventions: Genetic: Next generation sequencing (NGS)

INTERVENTIONS:
Genetic: Next generation sequencing (NGS) — NGS panel, whole exome / genome sequencing (WES/WGS), transcriptome analysis

SUMMARY:
The scientific aims of the project are to understand the genetic basis of Familial Hypercholesterolaemia (FH) in the Emirati population and estimate the overall prevalence of the disease. In addition, a clinical aim of the project is to explore the effectiveness of screening the relatives of individuals affected by FH and other lipid disorders ("cascade" screening) within Emirati families.

DETAILED DESCRIPTION:
Familial Hypercholesterolaemia is an inherited genetic disorder which causes elevated levels of low density lipoprotein (LDL) cholesterol in the blood. High LDL is a risk factor for with arterial disease and people with FH develop coronary artery disease (CAD) early in life. People with only one inherited copy of the defective gene usually develop CAD before the age of 60, whereas individuals who have inherited two copies usually die before the age of 30 from myocardial infarction ("heart attack") or sudden cardiac death. Coronary artery disease is a major cause of death and disability in the United Arab Emirates (UAE), and the medical costs associated with treating this condition are significant. Early identification and treatment of affected individuals can substantially postpone the onset of arterial disease and reduce the risk of mortality. In clinical practice, FH cases are usually identified by screening the relatives of people known to be affected.

Current study will focus on identifying individuals with high risk score for FH, based on the available medical records and laboratory information system (LIS). Furthermore, patients with history of premature ischaemic vascular disease and/or high readings for LDL-C will be approached and asked to participate.

The scientific aims of the study are:

* Identifying individuals with likelihood of FH diagnosis and confirming FH by genetic testing (applying Next Generation Sequencing NGS technology to analyse the genes already known and/or suspected to cause FH).
* Identifying novel FH genes and mutations in the Emirati population by performing whole exome and whole genome sequencing
* Validating positive genetic test results by performing mutational analysis on parental samples (if available)
* Introducing cascade screening on a clinical basis in order to identify affected relatives of those index individuals with a clinical diagnosis of FH
* Determining the prevalence of FH in the UAE
* Determining the short and the long-term clinical outcomes of FH in the UAE

It is expected that the cascade screening will provide additional clinical benefit to study participants and their families in terms of early identification and treatment where diagnosis could otherwise be missed. Early recognition and treatment in individuals with FH has been shown to reduce morbidity and mortality of affected individuals. The information gathered during this project will help introduce a cost-effective method for identifying people with dyslipidaemias and provide early intervention and management.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending Imperial College London Diabetes Centre
* Patients with hypercholesterolaemia
* Patients with possible evidence of known premature coronary heart disease (CHD)
* Patients (or parent/legal guardian if <18 years) willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Patients with no history of hypercholesterolaemia
* Patients or their legal guardian/legal representative who are unwilling or unable to give informed consent.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hypercholesterolaemia attending Imperial College London Diabetes Centre, UAE.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-17 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Next generation sequencing (NGS) | through study completion, an average of 2 year
  Identify individuals with likelihood of FH diagnosis and confirming FH by genetic testing (applying NGS technology to analyse the genes already known and/or suspected to cause FH).Identifying novel FH genes and mutations in the Emirati population by performing whole exome and whole genome sequencing (WES/WGS).

SECONDARY OUTCOMES:
Genetic test validation | through study completion, an average of 2 year
  Validating positive genetic test results by performing mutational analysis on parental samples (if available)
Cascade screening | through study completion, an average of 2 year
  Introduce cascade screening on a clinical basis in order to identify affected relatives of those index individuals with a clinical diagnosis of FH
Prevalence of FH | through study completion, an average of 2 year
  Determine the prevalence of FH in the UAE

CONTACTS AND LOCATIONS:
Overall Officials: Maha Barakat, PhD FRCP, Principal Investigator — Imperial College London Diabetes Centre
Locations (1):
- Imperial College London Diabetes Centre, Abu Dhabi, United Arab Emirates